CLINICAL TRIAL: NCT03809065
Title: Effects of Nitroglycerin Versus Labetalol on Tissue Perfusion During Deliberate Hypotension for Sinus Endoscopic Surgery.
Brief Title: Effects of Nitroglycerin Versus Labetalol on Tissue Perfusion During Deliberate Hypotension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Nassar,MD, Associate professor of Anesthesia, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: N53-2016
Record Dates: First submitted 2019-01-13; First posted 2019-01-18 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Tissue Perfusion; Deliberate Hypotension; Sinus Endoscopic Surgery
Keywords: Deliberate hypotension; Nitroglycerin; Labetalol; Peripheral perfusion
MeSH Terms: interventions — Nitroglycerin; Labetalol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group N (Experimental): Patients in this group will receive Nitroglycerin infusion for deliberate hypotension at a rate of 0.5-2 μg /kg/min .
  Interventions: Drug: Nitroglycerin
- group L (Active Comparator): Patients in this group will receive Labetalol infusion for deliberate hypotension at a rate of be 0.5-2 mg/kg/h .
  Interventions: Drug: Labetalol

INTERVENTIONS:
Drug: Nitroglycerin — Nitroglycerin is a direct vasodilator and its main action is through venodilation. Nitroglycerin will be diluted by adding 3 mL (3 mg) to 47 mL normal saline in a 50 mL syringe and will be infused after endotracheal intubation with a starting dose of 0.5 mL/Kg/ hr to have a starting dose of 0.5 μg/Kg/min. The rate of nitroglycerin infusion will be 0.5-2 μg /kg/min .The infusion rate will be finely adjusted to maintain MAP around 55-65mmHg or till reaching adequate surgical field {defined as surgical field score (SFS) <3}.
  Arms: group N
Drug: Labetalol — Labetalol is an α and β - adrenergic receptors competitive antagonist. Labetalol will be diluted by adding 10 mL (50 mg) to 40 mL normal saline in a 50 mL syringe and will be infused after endotracheal intubation with a starting dose of 0.5 mL/Kg/ hr. The rate of Labetalol infusion will be 0.5-2 mg/kg/h.The infusion rate will be finely adjusted to maintain MAP around 55-65mmHg or till reaching adequate surgical field {defined as surgical field score (SFS) <3}.
  Arms: group L

SUMMARY:
Deliberate hypotension is used to provide bloodless field during endoscopic sinus surgery; however, hypotension might impair perfusion of vital organs. The aim of this work is to compare the impact of nitroglycerin and labetalol on peripheral perfusion when used for induction of deliberate hypotension

DETAILED DESCRIPTION:
Hypotensive anesthesia is associated with the risk of reduced tissue perfusion. The usual target mean arterial pressure during deliberate hypotension is 50- 65 mmHg; however, the status of peripheral perfusion under this target is not well investigated. Nitroglycerin and Labetalol are commonly used drugs to achieve deliberate hypotension. Nitroglycerin is a direct vasodilator and its main action is through venodilation, while labetalol combines a selective α1 and non selective beta-adrenergic blocking activity. Both drugs were previously compared during deliberate hypotension with regard to surgical field quality and blood loss. No study to date compared the effects of both drugs on peripheral perfusion when used for induction of deliberate hypotension. The Peripheral Perfusion Index (PPI) is the ratio between pulsatile and non-pulsatile components of peripheral circulation. Measurement of PPI is based on analysis of the pulse oximetry signal. PPI showed increasing popularity as a non invasive monitor of peripheral perfusion. Serum lactate is another frequently used marker of global tissue perfusion.The aim of this study is to compare the influence of nitroglycerin and labetalol on tissue perfusion when used for induction of deliberate hypotension during FESS operations. Tissue perfusion will be evaluated using PPI and serum lactate as markers of peripheral and global tissue perfusion respectively.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female patients
* 18-45 years
* ASA physical status I-II
* scheduled for FESS operations

Exclusion Criteria:

* uncontrolled hypertension
* cerebrovascular disorders
* coagulation disorders
* cardiovascular diseases
* renal impairment
* liver impairment
* history of allergic reaction to any of the study medications

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-19 (Actual); Primary Completion 2019-05-25 (Actual); Study Completion 2019-05-25 (Actual)

PRIMARY OUTCOMES:
Peripheral perfusion index | 4 hours
  Peripheral perfusion index will be used as a marker of peripheral perfusion.

SECONDARY OUTCOMES:
Change in serum lactate concentration | Immediately before induction of anesthesia and after 60 minutes post recovery.
  Serum lactate concentration will be used as a marker of global tissue perfusion.Two samples will be obtained.
Total blood loss | from beginning of surgery till the end of the procedure
  Total blood loss will be measured from the suction device and gauzes that will be used to dry the surgical field.
Surgical field score (SFS) | from beginning of surgery till the end of the procedure.
  SFS ranges from 0 to 5 as follows: 0: No bleeding, 1: Slight bleeding-no suctioning of blood required, 2: Slight bleeding-occasional suctioning required. Surgical field not threatened. 3: Slight bleeding-frequent suctioning required. Bleeding threatens surgical field a few seconds after suction is removed, 4: Moderate bleeding-frequent suctioning required. Bleeding threatens surgical field directly after suction is removed, 5: Severe bleeding-constant suctioning required. Bleeding appears faster that can be removed by suction. Surgical field severely threatened and surgery not possible.
  Adequate surgical field is defined as SFS <3
Mean arterial blood pressure | 4 hours
  Target mean arterial pressure during deliberate hypotension will be 55-65mmHg
Heart rate | 4 hours
  Number of heart beats per minute

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Al Ainy, Cairo, Egypt

REFERENCES:
- [Derived] Zayed M, Nassar H, Hasanin A, Saleh AH, Hassan P, Saad D, Mahmoud S, Abo Bakr G, Fouad E, Saleh N, Ismail M, El-Hadi H. Effects of nitroglycerin versus labetalol on peripheral perfusion during deliberate hypotension for sinus endoscopic surgery: a randomized, controlled, double-blinded trial. BMC Anesthesiol. 2020 Apr 17;20(1):85. doi: 10.1186/s12871-020-01006-w. PMID 32303182